CLINICAL TRIAL: NCT02542007
Title: RECOVERY: A Prospective, Multi-center, Randomized Controlled Trial Evaluating the Safety and Efficacy of the Combo Bio-engineered Sirolimus-eluting Stent Versus the Nano Polymer-free Sirolimus-eluting Stent in the Treatment of Patients With de Novo Stenotic Lesions of Native Coronary Artery
Brief Title: Safety and Efficacy of the Combo Bio-engineered Sirolimus-eluting Stent Versus the Nano Polymer-free Sirolimus-eluting Stent in the Treatment of Patients With de Novo Stenotic Lesions
Acronym: RECOVERY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OrbusNeich (Industry)
Collaborators: CCRF Inc., Beijing, China (Industry); OrbusNeich Medical (Shenzhen), Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RECOVERY Combo 2015-01
Record Dates: First submitted 2015-09-01; First posted 2015-09-04 (Estimated); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Coronary Arteriosclerosis
Keywords: intracoronary stent; drug eluting stent; sirolimus; endothelial progenitor cells
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- OrbusNeich Combo stent™ (Experimental): The Combo Stent is composed of the OrbusNeich R stent™, with an abluminal coating of a bioabsorbable polymer matrix formulated with sirolimus for sustained release, and an anti-CD34 antibody cell capture coating on the luminal surface.
  Interventions: Device: OrbusNeich Combo stent™
- Nano Polymer-free sirolimus-eluting stent system (Active Comparator): The Nano polymer-free sirolimus-eluting stent produced by LePu medical.
  Interventions: Device: sirolimus-eluting stent system

INTERVENTIONS:
Device: OrbusNeich Combo stent™ — The Combo Stent is composed of the OrbusNeich R stent™, with an abluminal coating of a bioabsorbable polymer matrix formulated with sirolimus for sustained release, and an anti-CD34 antibody cell capture coating on the luminal surface.
  Arms: OrbusNeich Combo stent™
Device: sirolimus-eluting stent system
  Other Names: Nano Polymer-free sirolimus-eluting stent system
  Arms: Nano Polymer-free sirolimus-eluting stent system

SUMMARY:
To evaluate the safety, efficacy and deliverability of the Combo bio-engineered sirolimus-eluting stent versus the Nano polymer-free sirolimus- eluting stents in the treatment of patients with de novo stenotic lesions of native coronary artery.

DETAILED DESCRIPTION:
This is a prospective, multi-center, open-label, non-inferiority, randomized controlled trial which plans to enroll 436 subjects. All subjects enrolled will be randomly assigned to the test group (n=218) and the control group (n=218). Subjects in the test group and the control group will receive Combo stents and Nano stents respectively.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical evidence of asymptomatic or symptomatic ischemic heart disease, stable or unstable angina, old myocardial infarction;
* De novo lesions of native coronary arteries (lesions number ≤2);
* Target lesion located in one or two different vessels. The number of target lesions in one vessel shall be no more than one;
* Target vessel diameter between 2.5 and 4.0 mm by visual estimation. Target lesion length ≤ 32mm by visual estimation, which can be covered by one Combo stent with length 38mm or one Nano stent with length 36mm. It is suggested that the selected stent size should cover at least 2 mm (by visual estimation) of normal tissue on each side of the lesion;
* Target lesion diameter stenosis ≥ 70% by visual estimation;
* Each target lesion is permitted to implant only one stent at most, except bailout stent;
* Patients is eligible for PCI and is an acceptable candidate for CABG;
* Patients with left ventricular ejection fraction (LVEF) ≥40%;
* Patients who can understand the nature of the study, agree to participate and accept angiographic and clinical follow-up, and have provided written informed consent;

Exclusion Criteria:

* Patients with acute myocardial infarction (AMI) within one week;
* Chronic total occlusion lesion (TIMI 0 flow), Left main disease, Ostial lesion, and/or triple-vessel lesion that might require treatment, bifurcation lesions with a side branch diameter >2.5mm or graft lesions;
* Heavily calcified or tortuous lesions which cannot be successfully pre-dilated, and lesions which are not suitable for stent delivery and deployment;
* In-stent restenosis;
* Thrombotic lesion;
* Patients who had received any other stent in the past six months;
* Patients with acute or chronic renal dysfunction (defined as creatinine greater than 2.0 mg/dl);
* Patients with cardiogenic shock, acute infection, known bleeding or coagulation disorder, or with a history of active gastrointestinal bleeding, ulcer, cerebral hemorrhage or subarachnoid hemorrhage and stroke within 6 months;
* Patients who are allergic to aspirin, clopidogrel, ticagrelor, ticlopidine, heparin, contrast agent, sirolimus, stainless steel , polymer, or with contraindication to aspirin or clopidogrel or ticagrelor;
* Patients who had previously received murine therapeutic antibodies and exhibited sensitization through the production of HAMA;
* Patients with a life expectancy less than 1year;
* Patients who had participated in another investigational drug or device trial that has not completed the primary endpoint;
* Patient who has received any organ transplant or is on a waiting list for any organ transplant;
* Patient is in the opinion of the investigator, unable to comply with the requirements of the study protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Actual)
Dates: Start 2015-05; Primary Completion 2017-05-27 (Actual); Study Completion 2021-06-10 (Actual)

PRIMARY OUTCOMES:
In-segment late lumen loss (LLL) | 9 months post-procedure
  In-segment late lumen loss (LLL) refers to within the margins of the stent and 5 mm proximal and 5 mm distal to the stent.

SECONDARY OUTCOMES:
Device-oriented target lesion failure (TLF) | 30 days, 6 months, 12 months and annually up to 5 years
  The device-oriented target lesion failure (TLF) defined as a composite of cardiac death, target vessel myocardial infarction (MI), and ischemia-driven target lesion revascularization (i-TLR)
Patient-oriented composite endpoint | 30 days, 6 months, 12 months and annually up to 5 years
  The patient-oriented composite endpoint includes all-cause death, all MIs, or any revascularization
In-stent late lumen loss (LLL) | 9 months post-procedure
In-stent and In-segment binary restenosis (BR) | 9 months post-procedure
In-stent and In-segment minimal lumen diameter (MLD) | 9 months post-procedure
Definite and probable stent thrombosis (ST) | acute (0-24 hours), sub-acute (24 Hours to 30 Days), late (30 Days to 1 year) and very late (1 year to 5 years) period per Academic Research Consortium (ARC) definition criteria
  Definite and probable stent thrombosis (ST) in acute, sub-acute, late and very late period per Academic Research Consortium (ARC) definition criteria

CONTACTS AND LOCATIONS:
Overall Officials: Tao Ling, M.D., Principal Investigator — The First Affiliated Hospital of the Fourth Medical University; Xu Bo, M.D, Principal Investigator — The Secondary Affiliated Hospital of Harbin University
Locations (15):
- China (15):
  - Daqing General Oilfield Hospital, Daqing, Heilongjiang
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Nanjing First Hospital, Nanjing, Jiangsu
  - China Japan Union Hospital of Jilin University, Changchun, Jilin
  - The people Hospital of Liaoning Province, Shenyang, Liaoning
  - The Secondary Affiliated Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Kunming General Hospital of Chengdu Military region, Kunming, Yunnan
  - Beijing Chao Yang Hospital, Beijing
  - The Military General Hospital of Beijing PLA, Beijing
  - Bethune International Peace Hospital, Shijiazhuang
  - TEDA International Cardiovascular Hospital, Tianjin
  - Tianjin Medical University General Hospital, Tianjin
  - Tianjing Chest Hospital, Tianjing
  - The First Affiliated Hospital of the Fourth Military Medical University, Xi'an, Shanxi